CLINICAL TRIAL: NCT05250037
Title: The Longitudinal Impact of Respiratory Viruses on Bronchiolitis Obliterans Syndrome After Allogeneic Hematopoietic Cell Transplantation (The RV-BOS Study)
Status: Recruiting | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: RG1121806; NCI-2021-13375 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10767 (Other: Fred Hutch/University of Washington Cancer Consortium); R01HL161037 (NIH)
Record Dates: First submitted 2022-01-20; First posted 2022-02-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Bronchiolitis Obliterans Syndrome; Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Hematologic Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum, PBMC and nasal swabs.

GROUPS / COHORTS (1):
- Screening (spirometry measurements): Patients undergo home spirometry measurements with a portable handheld spirometer and complete questionnaires weekly, a nasal swab for viral polymerase chain reaction (PCR) surveillance every 4 weeks, and undergo blood collection and nasal swabs every 3 months for up to 2 years.
  Interventions: Procedure: Home spirometry; Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Home spirometry — Undergo spirometry measurements
  Other Names: SPIROMETRY
Procedure: Biospecimen Collection — Undergo nasal and/or oral swabs, and blood collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This observational trial studies whether respiratory viruses are the cause of lung disease (bronchiolitis obliterans syndrome [BOS] or graft-versus-host disease of the lung) and changes in lung function in patients who have received a donor stem cell transplant. Patients with chronic graft-versus-host disease (cGVHD) are at higher risk of developing BOS. Studies have also shown that patients who had a respiratory viral illness early after their transplant are at higher risk of developing lung problems later on. Patients who are at risk and who already have BOS might benefit from being monitored more closely. Spirometry is a way of assessing a patient's lung function and is often used to diagnose lung disease. Spirometry measured at home with a simple handheld device may reduce the burden of performing pulmonary function testing at a facility and potentially help patients get their lung disease diagnosed and treated sooner.

DETAILED DESCRIPTION:
OUTLINE:

This is an observational study.

Patients undergo home spirometry measurements with a portable handheld spirometer and complete questionnaires weekly, a nasal swab for viral polymerase chain reaction (PCR) surveillance every 4 weeks, and undergo blood collection and nasal swabs every 3 months for up to 2 years. (The minimum required follow-up is 1 year, but there is an optional 1 year extension period.)

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic HCT recipients with any indication, graft source, donor type, or conditioning regimen
* Age 8 and older
* COHORT 1 Inclusion criteria: One or more of the following clinical scenarios that encompass increased risk for BOS:

  1. A diagnosis of cGVHD as per NIH criteria through 5 years of diagnosis.

     i. New diagnosis of cGVHD within 3 months. This window may be extended by 30 days on a case-by-case basis.

     ii. A diagnosis of cGVHD ≥ 3 months ≤ 5 years with a new FEV1 decline of ≥10% in absolute compared with prior 2 years PFT.

     iii. A recent documented respiratory infection of any etiology that has been clinically managed and stabilized or improving as determined by a clinician, within 8 weeks.

     iv. Progression of flare of chronic GVHD requiring an alteration in therapy as determined by a clinician, within 3 months.
  2. At 'Day 80' evaluation. D80 designates posttransplant landmark, usually between 70-120 days, in which patients are evaluated for discharge back to community care. Patients with the following occurrences can be enrolled with 3 months of the Day 80 post-transplant evaluation.

     i. FEV1 decline of 10% in absolute values compared with pretransplant baseline. ii. Documented posttransplant RVI. iii. Lower respiratory tract disease (LRTD) of any etiology.
* COHORT 2 inclusion criteria: Newly diagnosed BOS within 6 weeks of clinical recognition. This may include the following scenarios:

  1. "Early BOS", ie patients with new airflow decline and obstruction, not yet meeting the FEV1 cut-off of < 75% predicted by FEV1, in the absence of other etiologies as determined by clinical investigations including chest imaging and microbiologic studies.
  2. NIH-defined BOS:

     i. FEV1 < 75% predicted, with a decline in absolute FEV1 > 10% compared to pretransplant baseline or within the prior 2 years. Absolute decline in FEV1 should remain >10% after bronchodilator response.

     ii. FEV1/FVC or FEV1/VC <0.7, or Lower Limit of Normal as per accepted reference standards. Reference standards may include National Health and Nutrition Examination Survey III or Global Lung Initiative.

     iii. Absence of an alternative diagnosis, including COPD exacerbation, asthma, and active respiratory tract infection, as determined by appropriate clinical investigations that may include chest imaging, microbiologic cultures, and/or bronchoscopy.

     iv. One of two supportive features of BOS:
     * a. Evidence of air trapping by PFTs: RV>120%, or elevated RV/TLC (>20% of predicted value)
     * b. High resolution chest CT with inspiratory and expiratory cuts that show findings that are consistent with small airways disease including (but not exclusive of) air trapping, bronchial wall thickening, or bronchiectasis.
  3. BOS with atypical spirometric pattern

     i. FEV1 <80%, with a preserved FEV1/FVC ratio (≥0.7) and TLC ≥80% in the absence of other clinically determined lung disease.
  4. Clinical or suspected diagnosis of BOS not otherwise meeting above criteria.
* Patient should have an Android or iOS-based smartphone with reliable access to Wi-Fi for data to be transmitted electronically. Android smartphones should have a software version of 4.0 or higher; iOS phones should have a version of 8.0 or higher.
* Patient should be willing and able to communicate electronically in English or Spanish.

Exclusion Criteria:

* Life expectancy < 2 years.
* Diagnosis of active hematologic relapse or malignancy requiring active treatment that will affect that patient's ability to comply with study procedures.
* Patient should not have a clinically acute active lower respiratory tract infection or a clinically acute active noninfectious respiratory condition (i.e. COPD exacerbation, pleural effusion) at the time of enrollment. However, patient may become eligible once these conditions have stabilized or resolved as noted above.
* Inability or unwillingness to perform the study procedures, most of which are performed at home.
* Lack of a personal iOS or Android smartphone.
* Inability or unwillingness to communicate electronically.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Allogeneic hematopoietic cell transplant recipients, age 8 and up.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of bronchiolitis obliterans syndrome (BOS) | Up to 2 years
  Diagnosed by National Institute of Health criteria or clinical diagnosis in the absence of alternative diagnosis.
Pulmonary impairment | Up to 2 years
  Defined by temporal decline in forced expiratory volume in the first second (FEV1) determined by assessment of spirometry data.

SECONDARY OUTCOMES:
Time from respiratory viral infection and chronic graft-versus-host disease to FEV1 decline | Up to 2 years
FEV1 (percent predicted) at clinical recognition of BOS | Up to 2 years
Incidence of asymptomatic and symptomatic viral infections | Up to 2 years
  Will be determined by the longitudinal follow-up of this observational study.
Incidence of late onset noninfectious pulmonary complications | Up to 2 years
  Will be determined by the longitudinal follow-up of this observational study. Follow-up of clinical encounters will provide an epidemiology of the incidence of noninfectious and infectious pulmonary complications.
Incidence of non-viral infectious pulmonary complications | Up to 2 years
  Will be determined by the longitudinal follow-up of this observational study. Follow-up of clinical encounters will provide an epidemiology of the incidence of noninfectious and infectious pulmonary complications.
Establishment of a biorepository that includes blood samples, respiratory viral samples, and nasal microbiome samples from patients with clinically recognized BOS | Up to 2 years
  The biorepository including self-collected samples will be catalogued and organized in a central location that can be easily accessed through a gatekeeper system.

CONTACTS AND LOCATIONS:
Overall Officials: Guang-Shing Cheng, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (4):
- United States (4):
  - Stanford Cancer Institute, Palo Alto, California
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No